CLINICAL TRIAL: NCT04873895
Title: Phase 1B Study of Hepatic Chemoembolization Plus Axitinib and Hydroxychlorquine for Liver-Dominant Metastatic Adenocarcinoma Of The Colon And Rectum
Brief Title: TACE Plus Axitinib and Hydroxychlorquine for Liver-Dominant Metastatic Colorectal Cancer (CRC)
Acronym: TACE-Ax-HCQ
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: failure to accrue
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC03221
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Neoplasms Malignant
Keywords: colorectal cancer; liver metastases
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Axitinib; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: single-center open-label Phase 1B trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TACE+axitinib+HCQ (Experimental): 2 weeks of axitinib 5mg BID and hydroxychloroquine 600 mg BID followed by lobar or segmental trans arterial chemoembolization monthly until the entire tumor burden is treated, then continue axitinib/HCQ until progression or intolerable toxicity.
  Interventions: Drug: Axitinib 5 MG; Drug: Hydroxychloroquine Pill; Procedure: trans arterial chemoembolization

INTERVENTIONS:
Drug: Axitinib 5 MG — axitinib 5 mg po BID until progression or intolerance
Drug: Hydroxychloroquine Pill — hydroxychloroquine 600 mg po BID until progression or intolerance
Procedure: trans arterial chemoembolization — segmental or lobar TACE at 4-8 week intervals until entire tummy burden is treated.

SUMMARY:
Liver metastases are a leading cause of death among patients with metastatic colorectal cancer. Duration of disease control is short following 2nd-line or later systemic therapy. Liver-directed therapy such as TACE has a higher response rate and improves progression-free survival (PFS), but the benefit is still limited. Cancer cells escape ischemic cell death via autophagy and hypoxia-inducible factor (HIF) activation. We hypothesize that blocking autophagy and the vascular endothelial growth factor (VEGF) pathway will improve both response and PFS following TACE.

DETAILED DESCRIPTION:
Subjects with liver-dominant colorectal cancer metastases failing at least one line of systemic therapy will receive 2 weeks of axitinib 5mg twice daily (BID) and HCQ 600 mg BID followed by lobar or segmental TACE monthly until the entire tumor burden is treated, then continue axitinib/HCQ until progression or intolerable toxicity. Response and hepatic progression-free survival (HPFS) will be assessed one month post-TACE, then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more.
2. Pathologically-verified diagnosis of colorectal adenocarcinoma.
3. Measurable metastasis to liver with at least one dimension ≥ 1.0 cm.
4. Liver dominant metastases as judged by multidisciplinary team consensus review of cross-sectional imaging of the chest, abdomen and pelvis.
5. At least 2 weeks must have elapsed from the last dose of chemotherapy before starting HCQ and at least 4 weeks must have elapsed from the last dose of VEGF/VEGFR therapy prior to starting axitinib.
6. Subjects must be at least 2 weeks beyond prior radiotherapy or surgery, and have recovered from all therapy associated toxicities.
7. Eastern Cooperative Oncology Group (ECOG) Performance status must be 0-1 (see Appendix II).
8. Absolute granulocyte count > 1,500/ul, platelet count > 75,000/ul, International Normalized Ratio (INR) < 1.6
9. Serum creatinine < 2.0 mg/dl; serum bilirubin < 2.0 mg/dl.
10. Urine protein:creatinine ratio < 1 or 24-hour urine protein < 1 gm/day
11. Liver function Child-Pugh A
12. Competent and willing to provide informed consent
13. Patients of reproductive potential agree to use approved contraceptive methods per section 5.4

Exclusion Criteria:

1. Contraindications to angiography and selective visceral catheterization:

   1. severe allergy or intolerance to contrast media not controllable with prophylaxis.
   2. bleeding diathesis not correctable by usual forms of therapy.
   3. severe peripheral vascular disease precluding catheterization.
2. Contraindications to hepatic artery embolization:

   1. high risk of hepatic failure, indicated by the constellation of greater than 50% liver replacement by tumor, lactate dehydrogenase (LDH) >425 mU/ml, aspartate aminotransferase (AST) >100mU/ml. and bilirubin >2 mg/dl.
   2. tumor volume >75% of total liver volume.
   3. portal vein occlusion without hepatopetal collateral flow demonstrated by angiography; or portal hypertension with hepatofugal flow.
   4. hepatic encephalopathy.
3. Prior hepatic arterial infusion chemotherapy or hepatic radiation therapy. Prior surgical resection or ablation of liver metastases is acceptable.
4. No more than two prior lines of systemic chemotherapy.
5. Pregnancy or lactation
6. Known allergic reactions to irinotecan, HCQ or axitinib
7. Allergy to contrast not mitigated by usual prophylaxis
8. Serious infection requiring intravenous therapy.
9. Known retinal disease
10. Poorly controlled hypertension, defined as a blood pressure > 150/100 at the time of enrollment. Patients with a preexisting hypertension must be on a stable anti-hypertensive regimen
11. History of abdominal fistula, gastrointestinal perforation, or serious non-healing wounds, ulcers, or bone fractures
12. Known New York Heart Association class II or greater congestive heart failure (defined as symptoms of fatigue, dyspnea, or other symptoms with ordinary physical activity)
13. Known untreated brain metastases. History of treated metastases off steroids allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Serious adverse event (SAE) rate | 12 months
  SAE is scored by CTCAE v5 (G3 or higher) and the 2017 revision of the Society of Interventional Radiology (SIR) Complications Classification categories 3-5.

SECONDARY OUTCOMES:
objective response rate in the liver | 3 months
  complete and partial response rate by RECIST and modified RECIST
Hepatic progression-free survival | 12 months
  Time from initiation of therapy to progression in the liver by RECIST, death from any cause, or last documented progression-free status.
Progression-free survival | 12 months
  Time from initiation of therapy to progression anywhere by RECIST, death from any cause, or last documented progression-free status.
Overall survival | 24 months
  Time from initiation of therapy to death or last follow-up alive
axitinib treatment intensity | 12 months
  Weeks on axitinib therapy multiplied by percentage of initially prescribed dose

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Soulen, MD, Principal Investigator — Abramson Cancer Center
Locations (1):
- Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiorentini G, Sarti D, Nani R, Aliberti C, Fiorentini C, Guadagni S. Updates of colorectal cancer liver metastases therapy: review on DEBIRI. Hepat Oncol. 2020 Jan 21;7(1):HEP16. doi: 10.2217/hep-2019-0010. PMID 32273974
- [Background] Gade TPF, Tucker E, Nakazawa MS, Hunt SJ, Wong W, Krock B, Weber CN, Nadolski GJ, Clark TWI, Soulen MC, Furth EE, Winkler JD, Amaravadi RK, Simon MC. Ischemia Induces Quiescence and Autophagy Dependence in Hepatocellular Carcinoma. Radiology. 2017 Jun;283(3):702-710. doi: 10.1148/radiol.2017160728. Epub 2017 Mar 2. PMID 28253108
- [Background] Fiorentini G, Sarti D, Nardella M, Inchingolo R, Nestola M, Rebonato A, Guadagni S. Chemoembolization Alone or Associated With Bevacizumab for Therapy of Colorectal Cancer Metastases: Preliminary Results of a Randomized Study. In Vivo. 2020 Mar-Apr;34(2):683-686. doi: 10.21873/invivo.11824. PMID 32111770
- [Background] Chan SL, Yeo W, Mo F, Chan AWH, Koh J, Li L, Hui EP, Chong CCN, Lai PBS, Mok TSK, Yu SCH. A phase 2 study of the efficacy and biomarker on the combination of transarterial chemoembolization and axitinib in the treatment of inoperable hepatocellular carcinoma. Cancer. 2017 Oct 15;123(20):3977-3985. doi: 10.1002/cncr.30825. Epub 2017 Jun 22. PMID 28640364